CLINICAL TRIAL: NCT02971605
Title: Measurement of Persisting Changes in Emotional Brain Functioning Produced by Psilocybin
Brief Title: Persisting Effects of Psilocybin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00102081; R03DA042336 (NIH)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): Participants will be administered a 25 mg/70 kg dose of psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 25 mg/70 kg Psilocybin

SUMMARY:
The proposed pilot study will assess whether ingestion of a classic hallucinogen (psilocybin) leads to changes in emotion processing and neural circuitry that may predict repeated self-administration of this drug and underlie an atypical mechanism of abuse liability, which may vitally contribute to the understanding of the potential for abuse and the underlying mechanisms supporting abuse of classic hallucinogens.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have at least a high-school level of education or equivalent, and be fluent in English
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of the drug session day. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on the session day.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine.
* Agree not to take any "as needed" medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Have limited lifetime use of hallucinogens

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrilation), artificial heart valve, or stroke in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including mono-amine oxidase inhibitors (MAOIs). For individuals who have intermittent or "as needed" use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table
* Current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Current or past history within the last 5 years of meeting DSM-5 criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine)
* Have a first or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or Bipolar I or II Disorder
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* Head trauma
* Claustrophobia incompatible with scanning
* Cardiac pacemaker
* Implanted cardiac defibrillator
* Aneurysm brain clip
* Inner ear implant
* Prior history as a metal worker and/or certain metallic objects in the body -- must complete magnetic resonance imaging (MRI) screening form and be approved by MRI technologist before each scan

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick S Barrett, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared with qualified scientists upon request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psilocybin
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Psilocybin
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Education Level [Count of Participants; unit: Participants]
  High School/GED | 1
  College | 4
  Post-Graduate | 8

OUTCOME MEASURES:

1. Primary Outcome: Amygdala Response to Stimuli in the Emotion Recognition Test
Description: Blood oxygenation level-dependent (BOLD) percent signal change in response to stimuli in the emotion recognition task was measured in the left and right amygdala.
Time Frame: 1 day pre (baseline), 1 week post, and 1 month post session
Measure: Mean (Standard Error); unit: BOLD percent signal change
Groups:
- Baseline: One day prior to psilocybin administration.
- 1-week Post Session: One week post psilocybin (25 mg/70 kg) administration.
- 1-month Post Session: One month post psilocybin (25 mg/70 kg) administration.
Arm/Group | Baseline | 1-week Post Session | 1-month Post Session
Number analyzed (Participants) | 12 | 12 | 12
BOLD percent signal change
  L Amygdala contrast: Happy | 0.835 (0.342) | -0.759 (0.63) | 0.619 (0.449)
  L Amygdala contrast: Sad | 0.503 (0.403) | -0.514 (0.635) | 0.999 (0.563)
  L Amygdala contrast: Fearful | 0.525 (0.421) | -0.928 (0.696) | 0.664 (0.584)
  L Amygdala contrast: Angry | 0.514 (0.357) | -0.881 (0.703) | 1.131 (0.569)
  L Amygdala contrast: Neutral | 0.794 (0.437) | -0.825 (0.572) | 1.098 (0.582)
  R Amygdala contrast: Happy | 0.938 (0.388) | -0.052 (0.431) | 0.749 (0.478)
  R Amygdala contrast: Sad | 0.927 (0.423) | 0.004 (0.37) | 0.816 (0.444)
  R Amygdala contrast: Fearful | 0.979 (0.424) | -0.254 (0.481) | 0.617 (0.563)
  R Amygdala contrast: Angry | 0.834 (0.449) | -0.028 (0.39) | 0.689 (0.454)
  R Amygdala contrast: Neutral | 1.081 (0.428) | -0.256 (0.358) | 0.719 (0.476)

2. Secondary Outcome: Change in Longitudinal Emotion and Mood Questionnaire Scores
Description: Participants were assessed on a variety of questionnaires that probed emotional functioning and mood state. Higher scores on each subscale are indicative of higher levels of each emotion/mood (e.g., low score on Depression (POMS) indicates low level of depressed mood).
  Depression Anxiety Stress Scale (DASS): Range 0-56 on all subscales
  Dispositional Positive Emotion Scale (DPES): Range 1-7 on all subscales
  Positive & Negative Affect Schedule Expanded (PANAS-X): Range 0-50 on all subscales
  Profile of Mood States (POMS): Ranges vary by subscale. Tension (0-36); Depression (0-60); Anger (0-48); Fatigue (0-28); Confusion (0-28); Vigor (0-36); Mood Disturbance (-36-168)
  State Trait Anxiety Inventory (STAI): Range 20-80 on all subscales
  Tellegen Absorption Scale (TAS): Range 0-34
  Big Five Inventory (BFI): Range 1-5 on all subscales
Time Frame: 1 day pre (baseline), 1 week post, and 1 month post session
Population: The Big Five Inventory (BFI) and the Tellegen Absorption Scale (TAS) were not administered at 1-week post, and were only administered at Baseline and 1-month post.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Baseline | 1-week Post Session | 1-month Post Session
Number analyzed (Participants) | 12 | 12 | 12
score on a scale
  Depression (DASS) | 1.82 (0.57) | 1.09 (0.73) | 1.64 (0.59)
  Anxiety (DASS) | 1.64 (1.07) | 1.64 (0.75) | 1.45 (0.90)
  Stress (DASS) | 4.91 (1.06) | 2.00 (0.60) | 3.27 (1.12)
  Joy (DPES) | 5.45 (0.21) | 6.02 (0.17) | 5.92 (0.21)
  Content (DPES) | 5.62 (0.24) | 6.27 (0.16) | 6.13 (0.23)
  Pride (DPES) | 5.42 (0.22) | 5.96 (0.14) | 5.95 (0.18)
  Love (DPES) | 5.61 (0.17) | 5.92 (0.25) | 5.98 (0.17)
  Compassion (DPES) | 5.75 (0.31) | 6.25 (0.26) | 6.00 (0.30)
  Amusement (DPES) | 5.02 (0.31) | 5.60 (0.32) | 5.71 (0.31)
  Awe (DPES) | 5.52 (0.26) | 6.06 (0.22) | 5.88 (0.24)
  Positive Affect (PANAS-X) | 38.18 (1.41) | 40.64 (1.28) | 40.18 (1.92)
  Negative Affect (PANAS-X) | 16.09 (1.00) | 12.36 (0.93) | 16.09 (0.80)
  Tension (POMS) | 4.82 (1.22) | 1.73 (0.49) | 3.82 (1.19)
  Depression (POMS) | 3.36 (0.81) | 0.55 (0.25) | 2.64 (1.03)
  Anger (POMS) | 4.91 (1.34) | 2.18 (0.58) | 4.64 (0.98)
  Fatigue (POMS) | 4.09 (1.37) | 2.27 (1.21) | 2.72 (1.06)
  Confusion (POMS) | 5.55 (1.19) | 4.27 (0.79) | 4.72 (1.21)
  Vigor (POMS) | 19.09 (1.35) | 21.45 (1.77) | 22.09 (2.15)
  Mood Disturbance (POMS) | 3.64 (5.67) | -10.5 (3.23) | -3.55 (6.19)
  State Anxiety (STAI) | 28.0 (2.41) | 22.82 (1.37) | 25.64 (2.56)
  Trait Anxiety (STAI) | 31.36 (1.91) | 28.55 (1.32) | 25.64 (27.55)
  Extraversion (BFI): number analyzed (Participants) | 12 | 0 | 12
  Extraversion (BFI) | 3.46 (0.190) |  | 3.69 (0.183)
  Agreeableness (BFI): number analyzed (Participants) | 12 | 0 | 12
  Agreeableness (BFI) | 4.43 (0.099) |  | 4.33 (0.117)
  Conscientiousness (BFI): number analyzed (Participants) | 12 | 0 | 12
  Conscientiousness (BFI) | 3.82 (0.172) |  | 3.98 (0.159)
  Neuroticism (BFI): number analyzed (Participants) | 12 | 0 | 12
  Neuroticism (BFI) | 1.82 (0.213) |  | 1.67 (0.175)
  Openness (BFI): number analyzed (Participants) | 12 | 0 | 12
  Openness (BFI) | 4.17 (0.129) |  | 4.22 (0.151)
  Absorption (TAS): number analyzed (Participants) | 12 | 0 | 12
  Absorption (TAS) | 0.98 (0.176) |  | 1.31 (0.233)

3. Secondary Outcome: Change in Emotional Functioning Task Accuracy
Description: These tasks measure emotional responding that may be altered by psilocybin.
  Emotional discrimination task: participants were presented with images of emotional facial expressions or shapes (control), and were instructed to discriminate between the images.
  Emotion recognition task: participants were presented images of actors and were asked to identify the emotional facial expression (happy, sad, fear, angry, neutral) of each actor.
  Emotional conflict Stroop task: participants were shown emotional facial expressions (targets) with emotional words overlain (distractors) and were asked to identify the valence of the facial expression, either positive or negative.
Time Frame: 1 day pre (baseline), 1 week post, and 1 month post session
Measure: Mean (Standard Error); unit: percentage of correct responses
Arm/Group | Baseline | 1-week Post Session | 1-month Post Session
Number analyzed (Participants) | 12 | 12 | 12
percentage of correct responses
  Emotion recognition task: Happy | 92.6 (2.7) | 95.8 (2.1) | 97.9 (1.5)
  Emotion recognition task: Sad | 95.7 (2.1) | 93.8 (2.5) | 94.8 (2.3)
  Emotion recognition task: Fearful | 100.0 (0.0) | 99.0 (1.0) | 97.9 (1.5)
  Emotion recognition task: Angry | 97.9 (1.5) | 95.8 (2.1) | 99.0 (1.0)
  Emotion recognition task: Neutral | 93.8 (2.5) | 96.9 (1.8) | 100.0 (0.0)
  Emotion discrimination: Shapes (Control) | 97.0 (1.0) | 97.0 (1.0) | 95.0 (1.3)
  Emotion discrimination: Faces | 87.1 (2.4) | 92.3 (1.8) | 93.2 (1.7)
  Emotional conflict Stroop: Congruent | 99.5 (0.3) | 99.8 (0.2) | 99.5 (0.3)
  Emotional conflict Stroop: Incongruent | 98.1 (0.7) | 97.9 (0.7) | 98.4 (0.6)

4. Secondary Outcome: Change in Emotional Functioning Tasks Response Time (Milliseconds)
Description: as for outcome 3
Time Frame: 1-day pre (baseline), 1-week post, 1-month post session
Measure: Mean (Standard Error); unit: milliseconds
Arm/Group | Baseline | 1-week Post Session | 1-month Post Session
Number analyzed (Participants) | 12 | 12 | 12
milliseconds
  Emotion recognition task: Happy | 1670 (59.5) | 1383 (41.2) | 1454 (45.6)
  Emotion recognition task: Sad | 1539 (53.0) | 1458 (45.6) | 1596 (56.8)
  Emotion recognition task: Fearful | 1061 (27.2) | 1045 (31.8) | 1130 (40.8)
  Emotion recognition task: Angry | 1380 (45.9) | 1193 (36.4) | 1310 (40.9)
  Emotion recognition task: Neutral | 1305 (49.1) | 1594 (49.2) | 1017 (33.4)
  Emotion discrimination task: Shapes | 977.0 (212.9) | 1697 (414.1) | 1735 (434.9)
  Emotion discrimination task: Faces | 1803 (51.1) | 1572 (41.1) | 1522 (35.3)
  Emotional conflict Stroop: Congruent | 613.5 (6.32) | 606.3 (5.88) | 603.2 (7.18)
  Emotional conflict Stroop: Incongruent | 641.3 (7.14) | 631.4 (7.03) | 614.1 (6.71)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from Screening to 1-month post psilocybin session (32-70 days).
Arm/Group | Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin (N=13)
Cardiac event (Cardiac disorders) | 2 (2) — Systolic blood pressure higher than 170 mmHg at session timepoint Diastolic blood pressure higher than 100 mmHg at session timepoint. Heart rate higher than 110 beats per minute (BPM) at session timepoint.
Thyroid hormone changes (Endocrine disorders) | 1 (1) — Change in thyroid-stimulating hormone (TSH) and T4 thyroid hormone levels

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT02971605/Prot_SAP_000.pdf